CLINICAL TRIAL: NCT06119100
Title: Characterization of STEnotic Lesion Type of Haemodialysis Arteriovenous Fistulae by Ultrasonography and Correlation With the Outcomes of Percutaneous Transluminal Angioplasty
Brief Title: Correlation of Ultrasonographic Lesion Type Characterization With Angioplasty Outcomes in Failing Dialysis AVFs
Acronym: STELA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Stavros Spiliopoulos, Associate Professor of Diagnostic and Interventional Radiology, Attikon Hospital
Other Study IDs: 77758
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Dialysis Access Malfunction
Keywords: angioplasty; autologous artriovenous fistula; dialysis; ultrasound; stenosis; stenosis type characterization
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound characterization of stenotic lesion type — Target lesion type will be classified as restrictive, hyperplastic or mixed using high frequency Duplex ultrasound, before the angioplasty procedure and at 6 months follow up.

SUMMARY:
The continuous increase in the incidence of end stage renal disease and hemodialysis patients, has raised the interest of the vascular access scientific community and many researchers are currently investigating the potential mechanisms of arteriovenous fistulas (AVF) dysfunction. Roy-Chaudhury et al. were the first to suggest neointimal hyperplasia (NIH) as the main reason of AVF dysfunction and vessel negative remodeling as another important factor. First, Yamamoto et al. described 3 stenotic lesions categories of arteriovenous grafts (AVG) observed by ultrasonography: 1. vascular constriction type, 2. neointimal hyperplasia type, 3. mixed type (constriction and neointimal hyperplastic type).

The main goals of this prospective observetional study are:

* The characterization of AVF stenotic lesions by ultrasonography
* The correlation of the stenotic lesion type with the outcomes of percutaneous transluminal angioplasty and the rate of reintervention.

DETAILED DESCRIPTION:
This is a prospective, observetional study designed to investigate the correlation of stenotic lesion type characterization (1. vascular constriction type, 2. neointimal hyperplasia type, 3. mixed type eg. constriction and neointimal hyperplastic type) using Duplex ultrasound, with the outcomes of high pressure plain balloon angioplasty. In total 200 patients with failing dialysis arteriovenoyus fistula (AVF) scheduled to undergo angioplasty of stenotic lesion(s) will be included. The study's primary endpoint will be the correlation between stenotic lesion type and target lesion re-intervention due to clinical recurrence at 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patiens with failing AVF scheduled to undergo fluoroscopically-guided high-pressure balloon angioplasty
* Signed study concent form

Exclusion Criteria:

* Patients undergoing dialysis via arteriovenous graft (AVG)
* Contraindications to angioplasty
* Immature AVF

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens between 18and 90 years of age, reffered due to failing AVF and scheduled to undergo fluoroscopically-guided, high-pressure balloon angioplasty of a significant stenosis within the dialysis access circuite.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation of target lesion reintervention (TLR) due to clinical recurrence and lesion type | 6 months
  The correlation of the speciific lesion type classified based on the pre-procedural ultrasonographic assessment and the target lesion reintervention rate due to clinical recurrence, will be investigated
Lesion characterization | Less than 48 hours before the procedure
  Lesion type will be classified as restrictive, hyperplastic or mixed based on the pre-procedural Duplex ultrasound assessment and the rates of each type will be recorded.

SECONDARY OUTCOMES:
Restenosis characterization post angioplasty | 6 months
  restenosis type will be classified as restrictive, hyperplastic or mixed based on the 6 months Duplex ultrasound assessment and the rates of each type will be recorded.
AVF survival | 6 months
  The overall AVF survival (secondary patency) will be recorded.
Binary restenosis rate | 6 months
  Binary (>50%) restenosis detected using Duplex ultrasound.
Periprocedural complication rate | Up to 48 hours post-procedure
  Procedure related complications rate

CONTACTS AND LOCATIONS:
Locations (1):
- "Attikon" University General Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided